CLINICAL TRIAL: NCT00408954
Title: A Multi Center Randomized Cross Over Double Blind Third Party Open Placebo Controlled Pilot Study to Assess the Urodynamic Effects of Modified Release UK-369,003 in Men With Lower Urinary Tract Symptoms.
Brief Title: Urodynamic Effects of UK-369,003 in Men With Lower Urinary Tract Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A3711045
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — 1-(6-ethoxy-5-(3-ethyl-6,7-dihydro-2-(2-methoxyethyl)-7-oxo-2H-pyrazolo(4,3-d)pyrimidin-5-yl)-3-pyridyl sulphonyl)-4-ethylpiperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: UK-369,003
- UK-369,003 (Active Comparator)
  Interventions: Drug: UK-369,003

INTERVENTIONS:
Drug: UK-369,003 — 100 mg MR tablet once daily for 2 weeks
  Arms: UK-369,003
Drug: UK-369,003 — UK-369,003-100 mg MR formulation for 2 weeks
  Arms: Placebo

SUMMARY:
This is a pilot study to generate hypotheses about the urodynamic effects of UK-369,003 in men with lower urinary tract symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, aged 40 years and above, with documented LUTS with an International Prostate Symptom Score (IPSS) ≥13.
* Clinical diagnosis of BPH
* Qmax 5 to 15 ml/sec with a voided volume of ≥150 ml
* Urodynamically defined bladder outlet obstruction

Exclusion Criteria:

* prostate cancer
* Post-void residual urine volume >200 ml
* Documented UTI
* History of relevant urological surgery

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
There is no specific primary endpoint for this study as it is not powered for that. It is mainly to generate hypotheses on the urodynamic effects of UK-369,003 in men with lower urinary tract symptoms. | Duration of study

SECONDARY OUTCOMES:
Maximum flow rate (Qmax) | Duration of study
Cystometric capacity | Duration of study
Post void residual volume (PVR) | Duration of study
Average flow rate (Qave) | Duration of study
Volume at first unstable contraction | Duration of study
Average detrusor pressure during micturition | Duration of study
Detrusor pressure at maximum flow rate (PdetQmax) | Duration of study
Bladder outlet obstruction index (BOOI) | Duration of study
Bladder contractility index (BCI) | Duration of study
Bladder voiding efficiency (BE) | Duration of study
Frequency of unstable contractions | Duration of study
International Prostate Symptom Score (IPSS) | Duration of study
Mean amplitude of unstable contractions | Duration of study
Patient Reported Treatment Impact (PRTI) | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Ústí nad Labem
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Nijmegen
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava, Slovakia
  - Pfizer Investigational Site, Martin, Slovakia
  - Pfizer Investigational Site, Trenčín, Slovakia
  - Pfizer Investigational Site, Košice

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3711045&StudyName=Urodynamic%20effects%20of%20UK-369%2C003%20in%20men%20with%20lower%20urinary%20tract%20symptoms.